CLINICAL TRIAL: NCT03336515
Title: Validity of a Vibrating Postural Device for the Treatment of Positional Obstructive Sleep Apnea (Postural)
Acronym: POSTURAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Araba (Other)
Collaborators: SIBEL SL (Unknown); Hospital Arnau de Vilanova (Other); Instituto de Salud Carlos III (Other Government); Instituto Vasco de Investigación Sanitaria (BIOEF) (Unknown)
Responsible Party: Principal Investigator, Joaquin Duran-Cantolla, MD, Principal Investigator. MD,PhD, Hospital Universitario Araba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014142
Record Dates: First submitted 2015-12-01; First posted 2017-11-08 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: OSA
Keywords: Positional Obstructive Sleep Apnea; Postural Device; Treatment
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A-General Recommendation (Other): General recommendation not sleeping in supine position without the postural device
  Interventions: Behavioral: Group A-General Recommendation
- Group B-Postural device no activated (Placebo Comparator): General recommendation not sleeping in supine position and the postural device without any activation (placebo)
  Interventions: Device: Group B-Postural device no activated
- Group C-Postural device activated (Experimental): General recommendation not sleeping in supine position and the postural device activated (intervention group).
  Interventions: Device: Group C-Postural device activated

INTERVENTIONS:
Device: Group C-Postural device activated — General recommendation not sleeping in supine position and the postural device activated (intervention group).
  Other Names: Intervention
  Arms: Group C-Postural device activated
Device: Group B-Postural device no activated — General recommendation not sleeping in supine position and the postural device without any activation (placebo)
  Other Names: Placebo
  Arms: Group B-Postural device no activated
Behavioral: Group A-General Recommendation — General recommendation not sleeping in supine position
  Other Names: Control
  Arms: Group A-General Recommendation

SUMMARY:
The objective of the study is validity of the effectiveness of a vibrating postural device in reduce the respiratory events (Apnea-Hypopnea Index-AHI) in patients with positional Obstructive Sleep Apnea (OSA).

DETAILED DESCRIPTION:
PURPOSE:

The objective of the study is validity of the effectiveness of a vibrating postural device in reduce the respiratory events (Apnea-Hypopnea Index-AHI) in patients with positional Obstructive Sleep Apnea (OSA).

The postural device is a vibratil device of 5x3 cm and a weight of about 30 grams integrating an accelerometer, a vibration and other sensors. The device is placed on the patient's forehead and when the device detects that the patient is in the supine position for 30 seconds or more, it starts a vibration, with increasing intensity, which ceases when the patient moves to lateral.

METHODOLOGY: DESIGN: A multicenter, randomized parallel study controlled by placebo. It will include patients with diagnosis of positional OSA in the Sleep Units of the Hospital Universitario Araba and Hospital Arnau de Vilanova de Lleida. These patients will be randomized to three groups: Group A: General recommendation not sleeping in supine position; Group B: General recommendation not sleeping in supine position and the device without any activation (placebo); Group C: General recommendation not sleeping in supine position and the device activated (intervention group).

Patients will undergo a basal conventional polysomnography (PSG) and after 12 weeks of treatment. In addition all patients will be visited at 1, 4, 8 and 12 weeks.

PRIMARY OUTCOME: Validity of the effectiveness of a vibrating postural device in reduce the respiratory events in patients with positional Obstructive Sleep Apnea . SECONDARY OUTCOMES: To determine the effectiveness of the device for: 1) To reduce the time spent in supine position; 2)To maintain the quantity and the quality of sleep; 3) The side effects ; 4) Reduction of snoring; 5) Cost-effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years old with diagnosis of positional OSA by PSG.
* Apnea-Hypopnea index (AHI) ≥ 5
* Apnea-Hypopnea index (AHI) in supine position doubling AHI in not supine position
* Time in supine position ≥ 20% total sleep time.
* Total sleep time at least 180 minutes
* Not received any treatment for OSA in the last four weeks before inclusion at the study (Except hygienic measures)
* Written informed consent signed.

Exclusion Criteria:

* Important problems of physical mobility
* Body mass index > 40kg/m²
* Presence of any previously diagnosed sleep disorders (narcolepsy, insomnia...) or difficulty in adopting a standard sleeping position
* Cognitive impairment, professional driver, use dangerous machinery, workers in three shifts, pregnant women or patients with severe disease.
* Patients with severe cardiovascular and/or respiratory comorbidity
* Excessive daytime sleepiness, Epworth scale >12
* Treatment with psychotropic drugs, central stimulant drugs, antidepressants, consumers of illegal drugs or consume > 80 grams of ethanol per day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI) | three month
  The effectiveness of the treatment will be measured by polysomnography (PSG), comparing the results of the basal PSG with the results of the final PSG (3 month), based on the results of the apnea hypopnea index (AHI).

SECONDARY OUTCOMES:
Reduce the time spent in supine position | three month
  To determine the effectiveness of the device for to reduce the time spent in supine position, measured by polysomnography, comparing the results of the basal PSG with the results of the final PSG (3 month).
Maintain the quantity and the quality of sleep | three month
  To determine the effectiveness of the device for to maintain the quantity and the quality of sleep, measured by polysomnography (PSG).
Side effects | three month
  To determine the side effects.
Reduction of snoring | three month
  To determine the effectiveness of the device for the reduction of snoring, measured by polysomnography (PSG).
Epworth Sleepiness Scale | at baseline and at three month of follow-up
  The Epworth Sleepiness Scale score (the sum of 8 items score, 0-3) can range from 0 to 24. Scores of 11-24 represent increasing levels of excessive daytime sleepiness.
Blood pressure | three month
  Blood pressure measurements: systolic blood pressure and diastolic blood pressure.
Anthropometric variables (Body mass index) | three month
  Body mass index
Quality of life (EuroQOL test) | at baseline and at three month of follow-up
  Evaluate by EuroQOL test, is a standardised measure of health status. Description of the state of health in five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression), each of wich is defined with three levels of severity, as measured by a Likert scale type(no problems, some problems and many problems or inability to activity).

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin Duran-Cantolla, MD, Principal Investigator — Hospital Universitario Araba; Jordi Rigau, Ing, Principal Investigator — Sibel SA
Locations (1):
- Hospital Universitario Araba, Vitoria-Gasteiz, Araba, Spain

REFERENCES:
- [Background] Duran J, Esnaola S, Rubio R, Iztueta A. Obstructive sleep apnea-hypopnea and related clinical features in a population-based sample of subjects aged 30 to 70 yr. Am J Respir Crit Care Med. 2001 Mar;163(3 Pt 1):685-9. doi: 10.1164/ajrccm.163.3.2005065. PMID 11254524
- [Background] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434
- [Background] Duran-Cantolla J, Mar J, de La Torre Munecas G, Rubio Aramendi R, Guerra L. [The availability in Spanish public hospitals of resources for diagnosing and treating sleep apnea-hypopnea syndrome]. Arch Bronconeumol. 2004 Jun;40(6):259-67. doi: 10.1016/s1579-2129(06)70096-9. Spanish. PMID 15161592
- [Background] Cartwright RD. Effect of sleep position on sleep apnea severity. Sleep. 1984;7(2):110-4. doi: 10.1093/sleep/7.2.110. PMID 6740055
- [Background] Oksenberg A, Silverberg DS, Arons E, Radwan H. Positional vs nonpositional obstructive sleep apnea patients: anthropomorphic, nocturnal polysomnographic, and multiple sleep latency test data. Chest. 1997 Sep;112(3):629-39. doi: 10.1378/chest.112.3.629. PMID 9315794
- [Background] Cartwright RD, Lloyd S, Lilie J, Kravitz H. Sleep position training as treatment for sleep apnea syndrome: a preliminary study. Sleep. 1985;8(2):87-94. doi: 10.1093/sleep/8.2.87. PMID 4012159
- [Background] Jokic R, Klimaszewski A, Crossley M, Sridhar G, Fitzpatrick MF. Positional treatment vs continuous positive airway pressure in patients with positional obstructive sleep apnea syndrome. Chest. 1999 Mar;115(3):771-81. doi: 10.1378/chest.115.3.771. PMID 10084491
- [Background] van Maanen JP, Richard W, Van Kesteren ER, Ravesloot MJ, Laman DM, Hilgevoord AA, de Vries N. Evaluation of a new simple treatment for positional sleep apnoea patients. J Sleep Res. 2012 Jun;21(3):322-9. doi: 10.1111/j.1365-2869.2011.00974.x. Epub 2011 Oct 22. PMID 22017727
- [Background] Ravesloot MJ, van Maanen JP, Dun L, de Vries N. The undervalued potential of positional therapy in position-dependent snoring and obstructive sleep apnea-a review of the literature. Sleep Breath. 2013 Mar;17(1):39-49. doi: 10.1007/s11325-012-0683-5. Epub 2012 Mar 24. PMID 22441662
- [Derived] Hidalgo-Armas L, Ingles S, Vaca R, Cordero-Guevara J, Duran-Carro J, Ullate J, Rigau J, Duran-Cantolla J; Spanish Sleep Network. Patient compliance and satisfaction with a new forehead device for positional obstructive sleep apnoea treatment: a post hoc analysis of a randomised controlled trial. BMJ Open Respir Res. 2023 Jun;10(1):e001503. doi: 10.1136/bmjresp-2022-001503. PMID 37349132
- [Derived] Hidalgo Armas L, Ingles S, Vaca R, Cordero-Guevara J, Duran Carro J, Ullate J, Barbe F, Duran-Cantolla J; Spanish Sleep Network. New forehead device in positional obstructive sleep apnoea: a randomised clinical trial. Thorax. 2021 Sep;76(9):930-938. doi: 10.1136/thoraxjnl-2020-216167. Epub 2021 Apr 22. PMID 33888576